CLINICAL TRIAL: NCT07397117
Title: Comparing Ultrasound-Guided Transgluteal Nerve Block to Standard Care for Emergency Department Patients With Low Back Pain and Sciatic Radiculopathy: A Randomized Controlled Trial
Brief Title: Comparing Ultrasound-Guided Transgluteal Nerve Block to Standard Care
Acronym: TGSNB vs SoC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-44506
Record Dates: First submitted 2026-01-25; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Sciatica Acute
Keywords: sciatica; sciatic back pain; lumbar radiculopathy; sciatic radiculopathy
MeSH Terms: conditions — Sciatica; Radiculopathy | interventions — Nerve Block; Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transgluteal sciatic nerve block (Experimental): Patients will receive an ultrasound-guided transgluteal sciatic nerve block with 10-20 mL of 0.2% ropivacaine injected around the affected sciatic nerve at the level of the greater trochanter.
  Interventions: Procedure: nerve block with ropivacaine
- Standard of care (Active Comparator): Standard ED analgesic management per departmental protocols (oral/IV NSAIDs, acetaminophen, opioids, muscle relaxants).
  Interventions: Other: Standard medical treatment

INTERVENTIONS:
Procedure: nerve block with ropivacaine — Ultrasound-guided transgluteal sciatic nerve block with 10-20 mL of 0.2% ropivacaine injected around the affected sciatic nerve at the level of the greater trochanter
  Arms: Transgluteal sciatic nerve block
Other: Standard medical treatment — Standard ED analgesic management per departmental protocols (oral/IV NSAIDs, acetaminophen, opioids, muscle relaxants).
  Arms: Standard of care

SUMMARY:
The goal of this clinical trial is to compare transgluteal sciatic nerve block to standard of care to treat sciatic back pain in adult patients who present to the emergency department.

The main question it aims to answer is: Is a transgluteal sciatic nerve block better than standard of care in improving pain in ER patients with sciatic back pain?

If there is a comparison group: Researchers will compare patients who receive transgluteal sciatic nerve blocks to patients who receive standard of care to see if pain scores improve in ER patients with sciatic back pain.

Participants will be randomized into the transgluteal sciatic nerve block group or the control group (standard of care). Participants will be asked to answer questions about their pain and will be asked to walk a timed short distance.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Presentation to ED with:
* Acute or acute-on-chronic pain consistent with sciatica, defined as unilateral lumbosacral radicular pain radiating from the lower back or gluteal region to the posterior leg, may extend distal to the knee.
* Pain score ≥ 5/10 on Numeric Rating Scale (NRS)

Exclusion Criteria:

* Known allergy to study medications (e.g., local anesthetics)
* Coagulopathy or current anticoagulation therapy
* Suspected or confirmed spinal infection, or tumor
* Neurological deficits (bowel or bladder dysfunction, leg weakness)
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Pain scores | 30 minutes after intervention, time of ED disposition (at decision point of admission to the hospital or discharge which can be up to 6 hours), 24 hours after ED visit, 48 hours after ED visit
  Patients in each group will be asked their pain score 30 minutes after their received intervention and at time of ED disposition (at decision point of admission to the hospital or discharge which can be up to 6 hours). Patients will then be contacted 24 and 48 hours after intervention to ask their pain score

SECONDARY OUTCOMES:
Ambulatory status | Before ED disposition, 24 and 48 hours after ED visit
  Before ED disposition, patients will be asked to perform another timed up and go (TUG) test. A patient rises from a chair, walks at a normal pace to a line (3 meters total), turns, walks back, and sits down. Patients will then be contacted 24 and 48 hours after intervention to ask about how their ambulatory status is.
ED Bouncback | 30 days after ED visit
  A chart review will be performed after 30 days to assess bounce-back rate

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Noble, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goldsmith AJ, Merz-Herrala J, Gullikson J, Selame LA, Cash RE, Martin D, Schwimmer H, Shokoohi H, Duggan NM, Nagdev A. The Efficacy of Ultrasound-Guided Transgluteal Sciatic Nerve Blocks for Sciatic Radiculopathy Pain in the Emergency Department: A Multicenter Prospective Study. J Am Coll Emerg Physicians Open. 2025 Apr 10;6(3):100137. doi: 10.1016/j.acepjo.2025.100137. eCollection 2025 Jun. PMID 40256350